CLINICAL TRIAL: NCT04524442
Title: A Multicenter, Open-label Post Authorization Safety Study to Evaluate the Effect of LysaKare® Infusion on Serum Potassium Levels in GEP-NET Patients Eligible for Lutathera® Treatment
Brief Title: Post-Authorization Safety Study (PASS) of LysaKare® in Adult Gastroenteropancreatic Neuroendocrine Tumor (GEP-NET) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAAA001A12401; 2019-004073-76 (EudraCT Number)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
Keywords: GEP-NET; Neuroendocrine tumors; NETs; carcinoid tumors; LysaKare; arginine/lysine; amino acid; Peptide Receptor Radionuclide Therapy; PRRT; Lutathera; Lutetium Lu 177 oxodotreotide; Lutetium Lu 177 dotatate
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors; Carcinoid Tumor | interventions — arginyllysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEP-NET (Experimental): One dose of arginine/lysine solution administered intravenously over a 4-hour period
  Interventions: Drug: arginine/lysine

INTERVENTIONS:
Drug: arginine/lysine — 1000 milliliters (mL) administered at a constant rate of 250 mL per hour
  Other Names: LysaKare

SUMMARY:
The purpose of the study was to evaluate the effect of arginine/lysine solution administration on serum potassium levels. A systematic assessment of serum potassium levels was performed during infusion and up to 24 hours post start of infusion compared to baseline.

DETAILED DESCRIPTION:
The study schedule for each patient consisted of a screening period followed by an infusion day with an optional overnight in-clinic stay, and a follow up call 48h post infusion.

Screening Phase:

At screening, patient eligibility was determined according to inclusion and exclusion criteria, with evaluation of patient's vital signs, ECG and laboratory parameters. The duration of screening could be as short as one day but could not exceed 7 days. Patients who showed potassium level > 6.0 mmol/L (> 5.5 mmol/L for Poland only) at screening could have their potassium level corrected and could be re-screened afterwards.

Treatment Phase:

Eligible patients were admitted to the in-clinic unit and dosed with arginine/lysine solution for infusion of 1,000 mL, which was administered intravenously over a period of 4 hours. Before the infusion (at 0 h time point), a set of baseline tests were performed. During and after the infusion, patient condition was monitored for evaluation of any adverse events. Only patients with a potassium level of ≤ 6 mmol/L at screening (> 5.5 mmol/L for Poland only) were allowed to be dosed. Potassium testing on the infusion day was performed at 0h (before the infusion), and at 2h, 4h, 6h, 8h, 12h, and 24h after the start of infusion. Vital signs and ECGs were taken as specified in the assessment schedule. All patients were monitored closely for signs and symptoms of hyperkalemia, e.g. dyspnoea, weakness, numbness, chest pain and cardiac manifestations (conduction abnormalities and cardiac arrhythmias). Other common adverse reactions during arginine/lysine solution administration are nausea and vomiting. Before the start of arginine/lysine solution infusion, an intravenous bolus of an anti-emetic was given. The choice of anti-emetic drugs was at the discretion of the physician.

Follow-up Phase:

All patients were called for a safety follow-up in 48 hours after dosing. Patients were not scheduled to receive repeat dosing with arginine/lysine solution as concomitant medication with Lutathera® within 7 days of the arginine/lysine solution infusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with somatostatin receptor positive gastroenteropancreatic neuroendocrine tumours (GEP-NETs), who are eligible for the treatment with Lutathera as per Lutathera label indication.
* Patients who have provided a signed informed consent form to participate in the study, obtained prior to the start of any protocol related procedures.

Exclusion Criteria:

* Pre-existing hyperkalemia (>6.0 mmol/L at screening) if not adequately corrected before starting the LysaKare (arginine/lysine) infusion. For Poland only, pre-existing hyperkalemia (> 5.5 mmol/L at screening) if not adequately corrected before starting the LysaKare (arginine/lysine) infusion.
* Instances when Lutathera is not recommended per the Lutathera Summary of Product Characteristics (SmPC).
* Pregnancy or lactation, positive pregnancy test at screening or pre-dose based on the contraindication for Lutathera.
* Any significant medical or social condition which may interfere with the subject's ability to comply with the study visit schedule or the study assessments.
* Patients who have received any investigational agent within the last 30 days.
* Patients that have received a dose of Lutathera prior to the screening visit or are scheduled for Peptide Receptor Repeat (PRRT) treatment within 7 days of the study infusion of arginine/lysine solution.
* Other protocol-defined exclusion criteria may apply.

Exclusion Criteria (Poland Only):

- Pre-existing hyperkalemia (> 5.5 mmol/L at screening) if not adequately corrected before starting the arginine/lysine solution infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Istituto Europeo di Oncologia, Milan, MI, Italy
- Erasmus University Medical Center, Rotterdam, Gelderland, Netherlands
- Gammed-Centrum Diagnostyczno-Lecznicze, Warsaw, Poland
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Royal Surrey Country Hospital, Guildford
  - Liverpool Royal Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants were enrolled in 7 centers in 4 countries.
Pre-assignment Details: The study schedule for each participant consisted of a screening period followed by an infusion day with an optional overnight in-clinic stay, and a follow-up call.
Period: Overall Study
Arm/Group | GEP-NET
Started | 42
Treated | 41
Not Treated | 1
Post-treatment Follow-up Phase (48 Hrs Post-infusion) | 40
Completed | 41
Not Completed | 1
Not completed — Subject Decision | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: The Safety Set (SAF) comprises all subjects who received any administration of the LysaKare infusion in the study.
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38
  Black or African American | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Serum Potassium Levels Over 24 Hours
Description: Serum potassium levels at each collection time point will be measured at local laboratories of study sites using validated methods. The potassium concentration results will be summarized descriptively and will include mean change, maximum change, time to the maximum change, and the overall dynamics of the potassium concentration curve during and after the arginine/lysine infusion.
Time Frame: Day 0/Infusion Day (Hour 0, Hour 2, Hour 4, Hour 6, Hour 8, Hour 12, Hour 24)
Population: Evaluable Set: The Evaluable Set comprises all subjects who received any volume of the LysaKare infusion and provided both pre-dose and at least one post-dose (between 4 and 8 hours) potassium levels measured from serum.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GEP-NET
Number analyzed (Participants) | 25
mmol/L
  Pre-dose (hour 0) | 4.3 (0.397)
  Change from Baseline (BL) to Hour 2: number analyzed (Participants) | 23
  Change from Baseline (BL) to Hour 2 | 0.25 (0.452)
  Change from Baseline (BL) to Hour 4 | 0.60 (0.666)
  Change from Baseline (BL) to Hour 6 | 0.49 (0.602)
  Change from Baseline (BL) to Hour 8 | 0.38 (0.487)
  Change from Baseline (BL) to Hour 12: number analyzed (Participants) | 24
  Change from Baseline (BL) to Hour 12 | 0.24 (0.557)
  Change from Baseline (BL) to Hour 24 | 0.07 (0.396)

2. Secondary Outcome: Percentage of Participants With Treatment Adverse Events (AEs) & Serious Adverse Events (SAEs)
Description: Safety measured by the percentage of participants with treatment emergent adverse events (starting from the signing of the ICF until the end of the follow-up call (48 hours after infusion).
Time Frame: Day 0/Infusion Day up to 48 hours post infusion
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants
  Adverse Event (AEs) | 11
  Treatment-related AEs | 6
  Serious Adverse Events (SAEs) | 0
  Fatal SAEs | 0
  AEs leading to discontinuation | 0
  AEs leading to Interrruption | 0
  AEs requiring additional therapy | 5
  Treatment related AEs req. additional therapy | 3

3. Secondary Outcome: Number of Participants With Notable Changes in Vital Signs
Description: Safety measured by the notable post-baseline changes in vital signs: (systolic blood pressure, diastolic blood pressure, pulse rate & weight) compared to baseline.
Time Frame: Day 0/Infusion Day (0, 2, 4, 6, 8, 12 and 24 hours)
Population: The Safety Set (SAF) comprises all subjects who received any administration of the LysaKare infusion in the study.
Measure: Number; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants
  Systolic blood pressure (mmHg): ≥180 with increase from baseline of ≥20 | 0
  Systolic blood pressure (mmHg): ≤ 90 with decrease from baseline of ≥20 | 0
  Diastolic blood pressure (mmHg): ≥105 with increase from baseline of ≥15 | 0
  Diastolic blood pressure (mmHg): ≤ 50 with decrease from baseline of ≥15 | 0
  Pulse rate (bpm): ≥100 with increase from baseline of >25% | 0
  Pulse rate (bpm): ≤ 50 with decrease from baseline of > 25% | 0
  Weight (kg): increase ≥10% from Baseline | 0
  Weight (kg): decrease > 10% from Baseline | 0

4. Secondary Outcome: Number of Participants With Notable Changes in Electrocardiogram (ECG)
Description: Safety measured by the notable post-baseline changes in ECG values compared to baseline PR, QRS, QT, QTcF, and RR intervals were obtained from 12-lead ECGs for each subject during the study
Time Frame: Day 0/Infusion Day (0, 4, 8 and 24 hours)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants
  QTcF (ms): Increase >30 to ≤ 60 ms | 7
  QTcF (ms): Increase >60 ms | 0
  QTcF (ms): New >450 to ≤ 480 ms: number analyzed (Participants) | 39
  QTcF (ms): New >450 to ≤ 480 ms | 7
  QTcF (ms): New >480 to ≤ 500 ms | 0
  QTcF (ms); New >500 ms | 0
  QT (ms): Increase >30 to ≤ 60 ms | 9
  QT (ms): Increase >60 ms | 2
  QT (ms): New >450 to ≤ 480 ms: number analyzed (Participants) | 39
  QT (ms): New >450 to ≤ 480 ms | 6
  QT (ms): New >480 to ≤ 500 ms | 1
  QT (ms): New >500 ms | 0
  PR (ms): Increase >25% and PR >200 ms: number analyzed (Participants) | 29
  PR (ms): Increase >25% and PR >200 ms | 1
  PR (ms): New PR >200 ms: number analyzed (Participants) | 29
  PR (ms): New PR >200 ms | 6
  QRS (ms): Increase >25% and QRS >120 ms | 2
  QRS (ms): New QRS >120 ms | 2
  HR (bpm): Increase >25% and HR >100 bpm | 0
  HR (bpm): Decrease >25% and HR <50 bpm | 0

5. Secondary Outcome: Number of Participants With Notable Changes in Hematology Parameters
Description: Safety measured by the notable post-baseline changes in Hematology parameters compared to baseline as represented by Shift tables based on common toxicity criteria (CTC) grades. Each participant was counted only for the worst grade observed post-baseline. Notable change is the shift to higher grades from baseline.
Time Frame: Day 0/Infusion Day (0 and 24 hours)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants | 0

6. Secondary Outcome: Number of Participants With Notable Changes in Chemistry Parameters
Description: Safety measured by the notable post-baseline changes in Chemistry parameters compared to baseline. Each participant was counted only for the worst grade observed post-baseline. Notable change is the shift to higher grades from baseline.
  Key shifts were in the following parameters: creatinine, lactate dehydrogenase and creatinine clearance.
Time Frame: Day 0/Infusion Day (0 and 24 hours)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants
  Creatinine (increase) | 4
  Lactate dehydrogenase (increase) | 3
  Creatinine clearance (decrease) | 4

7. Secondary Outcome: Number of Participants With Notable Changes in Electrolyte Parameters
Description: Safety measured by the notable post-baseline changes in Electrolyte parameters compared to baseline. Each participant was counted only for the worst grade observed post-baseline. Notable change is the shift to higher grades from baseline.
Time Frame: Day 0/Infusion Day (0, 2, 4, 6, 8, 12 and 24 hours)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
Participants
  For Potassium (increase) | 7
  For sodium (decrease) | 12

8. Secondary Outcome: Mean Change From Baseline in Blood Gas Parameter, pH, Over 24 Hours
Description: Safety measured by the mean changes in blood gas compared to baseline. Blood gas parameter: pH.
Time Frame: Day 0/Infusion Day (0, 2, 4, 6, 8, 12 and 24 hours)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
unitless
  Day 0/Infusion Day (Pre-dose) (hour 0): number analyzed (Participants) | 36
  Day 0/Infusion Day (Pre-dose) (hour 0) | 7.35 (0.046)
  Change from Baseline (BL) to Hour 2: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 2 | -0.03 (0.046)
  Change from Baseline (BL) to Hour 4: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 4 | -0.06 (0.055)
  Change from Baseline (BL) to Hour 6: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 6 | -0.05 (0.051)
  Change from Baseline (BL) to Hour 8: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 8 | -0.05 (0.056)
  Change from Baseline (BL) to Hour 12: number analyzed (Participants) | 33
  Change from Baseline (BL) to Hour 12 | -0.03 (0.054)
  Change from Baseline (BL) to Hour 24: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 24 | -0.04 (0.051)

9. Secondary Outcome: Mean Change From Baseline in Blood Gas Parameter, Lactic Acid, Over 24 Hours
Description: Safety measured by the mean changes in blood gas compared to baseline. Blood gas parameter: Lactic Acid
Time Frame: Day 0/Infusion Day (0, 2, 4, 6, 8, 12 and 24 hours)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
mmol/L
  Day 0/Infusion Day (Pre-dose) (hour 0): number analyzed (Participants) | 35
  Day 0/Infusion Day (Pre-dose) (hour 0) | 1.40 (0.604)
  Change from Baseline (BL) to Hour 2: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 2 | -0.07 (0.671)
  Change from Baseline (BL) to Hour 4: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 4 | -0.23 (0.523)
  Change from Baseline (BL) to Hour 6: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 6 | -0.26 (0.546)
  Change from Baseline (BL) to Hour 8: number analyzed (Participants) | 33
  Change from Baseline (BL) to Hour 8 | -0.19 (0.465)
  Change from Baseline (BL) to Hour 12: number analyzed (Participants) | 33
  Change from Baseline (BL) to Hour 12 | -0.21 (0.657)
  Change from Baseline (BL) to Hour 24: number analyzed (Participants) | 34
  Change from Baseline (BL) to Hour 24 | -0.16 (0.650)

10. Secondary Outcome: Mean Change From Baseline in Blood Gas Parameter, Partial Pressure Carbon Dioxide, Over 24 Hours
Description: Safety measured by the mean changes in blood gas compared to baseline. Blood gas parameter: Partial Pressure Carbon Dioxide.
Time Frame: Day 0/Infusion Day (0, 2, 4, 6, 8, 12 and 24 hours)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GEP-NET
Number analyzed (Participants) | 41
mmHg
  Day 0/Infusion Day (Pre-dose) (hour 0): number analyzed (Participants) | 36
  Day 0/Infusion Day (Pre-dose) (hour 0) | 50.53 (8.712)
  Change from Baseline (BL) to Hour 2: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 2 | -1.08 (6.670)
  Change from Baseline (BL) to Hour 4: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 4 | -2.44 (8.717)
  Change from Baseline (BL) to Hour 6: number analyzed (Participants) | 36
  Change from Baseline (BL) to Hour 6 | -4.90 (8.507)
  Change from Baseline (BL) to Hour 8: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 8 | -4.87 (8.399)
  Change from Baseline (BL) to Hour 12: number analyzed (Participants) | 33
  Change from Baseline (BL) to Hour 12 | -5.71 (8.002)
  Change from Baseline (BL) to Hour 24: number analyzed (Participants) | 35
  Change from Baseline (BL) to Hour 24 | -2.54 (8.242)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the administration of the study treatment up to 48 hours in addition to the infusion time, an average of 52 hours total.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up.
Groups:
- All Participants: All participants enrolled in the study who received one dose of arginine/lysine solution administered intravenously over a 4-hour period
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 11/41
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=41)
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04524442/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04524442/SAP_001.pdf